CLINICAL TRIAL: NCT01336218
Title: An Open-Label, Non-Randomized, 2-Period, Single Center Study to Assess the Single Dose Pharmacokinetics of R406 in Healthy Subjects When Fostamatinib 150 mg is Administered Alone and in Combination With Rifampicin
Brief Title: Effects of Administration of Fostamatinib on Blood Concentrations of Rifampicin in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Kelli Craven, MD, PI, Quintiles, Overland Park, volunteer recruitment
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D4300C00015
Record Dates: First submitted 2011-04-14; First posted 2011-04-15 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Rheumatoid Arthritis; Healthy Volunteers
Keywords: Phase 1; healthy volunteers; Rheumatoid arthritis; RA; Fostamatinib; Rifampicin; drug-drug interaction; Pharmacokinetics; Amount of Rifampicin in blood
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — fostamatinib; Rifampin

ARMS (2):
- 1 (Experimental): Fostamatinib
  Interventions: Drug: fostamatinib
- 2 (Experimental): Rifampicin
  Interventions: Drug: fostamatinib; Drug: rifampicin

INTERVENTIONS:
Drug: fostamatinib — oral tablets, 150mg (3 X 50mg) single dose per period
Drug: rifampicin — oral tablets, 600mg (2 X 300mg) 8 doses over 8 days
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the drug interaction between fostamatinib and rifampicin by comparing the safety, tolerability and plasma concentration of fostamatinib when administered alone and with rifampicin in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Males or females aged 18 to 55 years (inclusive)
* Minimum weight of 50 kg and a body mass index (BMI) of 18 to 35 kg/m2 (inclusive)
* Female subjects must have a negative pregnancy test at screening and admission of each treatment period, must not be lactating, and must be of non-childbearing potential

Exclusion Criteria:

* History or presence of gastrointestinal, hepatic or renal disease (except for cholecystectomy)
* Any clinically significant illness, medical or surgical procedure, or trauma within 4 weeks before Period 1 Day 1
* Subjects who smoke more than 5 cigarettes or the equivalent in tobacco per day
* Absolute neutrophil count of less than 2500/mm3 or 2.5 x 109/L
* Any previous treatment with fostamatinib

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2011-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To assess the pharmacokinetics of R406 in healthy subjects when a single dose of fostamatinib is administered alone and in combination with rifampicin. AUC and Cmax will be measured | Period 1: Day 1 to 96 hours post-dose Period 2: Day 6 to 96 hours post-dose

SECONDARY OUTCOMES:
To assess the pharmacokinetics of R406 in healthy subjects when a single dose of fostamatinib is administered alone and in combination with rifampicin. AUC (0-t), terminal half life, and tmax will be measured | Period 1: Day 1 to 96 hours post-dose Period 2: Day 6 to 96 hours post-dose
To examine the safety and tolerability of fostamatinib in combination with rifampicin. | From screening, Day 1 - Day 25, up to follow up visit
  Assessments include: Adverse events, laboratory assessments, vital signs, physical examination and 12-lead electrocardiogram. Absolute values and change in baseline for any of these parameters will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Overland Park, Kansas, United States